CLINICAL TRIAL: NCT07302555
Title: Outcomes of Patients Over 75 Years of Age Who Consulted the Emergency Department for a Medical Problem, Depending on Their Direct Admission to a Medical Ward Versus Prior Hospitalization in the Short-Stay Unit (UHCD).
Brief Title: Outcomes of Patients Over 75 Years of Age Who Consulted the Emergency Department for a Medical Problem
Acronym: GERIA-UH
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9452
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Medical Problem
Keywords: Acute medical problem; Patient over 75 years of age

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The increasing activity of emergency departments, coupled with a decrease in the number of hospital beds, is leading to operational changes, of which the Short-Stay Unit (UHCD) is one example. Initially designed for stays of less than 24 hours, it now finds itself providing supplementary hospitalization for downstream services, which is detrimental to the most vulnerable elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 75 years
* Patient admitted to the Strasbourg Emergency Department (Hautepierre and NHC) during 2019 for an acute medical problem
* Patient with an indication for hospitalization in a conventional medical ward

Exclusion Criteria:

* Patient who died during their visit to the Emergency Department prior to hospitalization
* Patient admitted for a scheduled hospitalization
* Patient not requiring hospitalization in a conventional medical ward (either discharged home after the Emergency Department visit or admitted to intensive care)
* Patient admitted to the Emergency Department for a surgical condition

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Patient aged ≥ 75 years admitted to the Strasbourg Emergency Department (Hautepierre and NHC) during 2019 for an acute medical problem
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
3-month mortality rate depending on whether or not they were hospitalized in the UHCD. | 3-month mortality rate after hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Soins de Soins Médicaux et de Réadaptation - Réanimation - CHU de Strasbourg - France, Strasbourg, France